CLINICAL TRIAL: NCT06254430
Title: Effects of Erector Spina Plan Block and Epidural Analgesia in Whipple Surgery
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Ayça Özcan, Principal Investigator, Ankara City Hospital Bilkent
Other Study IDs: E2-22-1596
Record Dates: First submitted 2023-12-19; First posted 2024-02-12 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Epidural analgesia: The patients were fasted for 8 hours before the operation without premedication. The patient was taken to the operation room. In all cases, a vein on the back of the hand was cannulated for peripheral venous catheter was cannulated from the back of the hand. Standard monitoring was applied.
  In the epidural group, 42 patients received a standard 18 G injection at the appropriate level between T8 and T10. The epidural space was entered by loss of resistance method with touchy needle. 15 µg in 3 mL saline The test dose was administered by administering epinephrine. Then the epidural catheter was inserted towards the cranium. was advanced five cm. Bupivacaine 0.25% was started as infusion through the catheter.
  Since the mean arterial pressure dropped below 60 mm/hg in 5 patients, epidural infusion was stopped and inotropic treatment was started.
- Erector Spina Plan(ESP) Block: Esp group included 28 patients in the preoperative operating theatre between T8 and T10 1 hour before the operation.
  level, the USG (ultrasonography) probe is placed in the midline in the cephalocaudal direction and then the USG (ultrasonography) probe is placed approximately 3 cm laterally over the transverse processes and transverse with the erector spinae muscle 0.25 % bupivacaine 20 cc each in the fascial plane between the processes bilateral thoracic erector spina block and then 50 mg dexketoprofen before surgery implemented.

SUMMARY:
Pancreatic surgery is generally a high-risk and difficult to manage perioperatively.

surgery. In pancreatic surgery, in addition to general anaesthesia, central blocks for analgesia and peripheral blocks are also preferred. In this study, in patients undergoing whipple surgery epidural and erector spina plan block (ESP) may cause intraoperative and postoperative pain, renal functions and haemodynamic variables.

DETAILED DESCRIPTION:
Pancreatic surgery and anaesthetic management is a difficult operation due to the anatomical location and function of the pancreas. Thoracic epidural anaesthesia/analgesia (TEA) in addition to general anaesthesia in upper abdominal surgeries such as pancreas, liver and stomach.Thoracic epidural analgesia (TEA) is the most widely used gold standard in this type of surgery.

TEA may cause haemodynamic changes in patients due to decreased sympathetic tone due to sympathetic nerve blockade. In elderly patients, bradycardia and hypotension is observed more frequently. Cardiovascular response decreases with age due to decreased cardiac reserve and deterioration of the autonomic nervous system and arteriolar structure. This can lead to this is because more segments are blocked than in younger patients. Pain control with thoracic epidural will provide pulmonary rehabilitation and rapid mobilisation. Accordingly, thromboembolic events, atelectasis and pulmonary infections are prevented. However, it has important unwanted side effects such as hypotension, dural puncture and contralateral block. All these disadvantages of TEA has increased interest in alternatives. Peripheral regional anaesthesia techniques have become more popular as a component of multimodal analgesia to avoid complications associated with epidural analgesia.

In 2016, ESP block, which is an ultrasound-controlled fascial plane block, was described. ESP block is considered to be an easier, effective and safer alternative to epidural and paravertebral blocks. The mechanism of action of ESP involves blockade of both dorsal and ventral branches, resulting in somatic and visceral analgesia.

Intraoperative and postoperative renal function may be impaired in upper abdominal surgeries. Acute kidney injury (AKI) is an important cause of postoperative mortality and morbidity. The most serious adverse factor is both surgical and anaesthesia-related AKI.

hypotension that may develop. The duties of the anaesthesiologist include maintaining perioperative renal function, predetermining the risk of AKI and taking necessary precautions. Considering the data in the literature, postoperative AKI Recent studies have shown that there is a link between inflammation and cancer. Studies reveal a relationship between cytokine and chemokine production and tumour growth, angiogenesis and metastatic capacity. Inflammatory cells and substances produced by inflammation affect cells in the peripheral blood. Platelets promote extravasation of circulating tumour cells. Neutrophils can also promote tumour adhesion and seeding by secreting growth factors into the peripheral circulation. However, lymphocytes can exert anti-tumour effects by inhibiting the proliferation and migration of tumour cells. From this point of view, SII (Systemic inflammation index) is a new prognostic factor obtained by measuring the number and ratio of neutrophils, platelets and lymphocytes in the peripheral blood of many tumours.

In this study, the effects of epidural analgesia and ESP block on intraoperative opioid requirement and postoperative pain scores, as well as perioperative renal parameters, haemodynamic data and SII (Systemic inflammation index) were investigated and the alternative of ESP block to epidural analgesia was investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing whipple surgery,
* ASA (The American Society of Anesthesiologists) I-III risk grup
* Between the ages of 18-80

Exclusion Criteria:

* Those who do not accept the transaction,
* Serious cardiovascular disease,
* Those for whom epidural anesthesia and peripheral blocks are contraindicated,
* Those who have had spinal surgery,
* Those who are allergic to one of the local anesthetics to be used,
* Those whose hemoglobin value is below 10 g/dl) disease,
* Those with drug and alcohol addiction,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who will have whipple surgery operation under general anesthesia in Ankara Bilkent City Hospital Operating Room,between the ages of 18-80,both genders and in the ASA (The American Society of Anesthesiologists) 1,2,3 risk grup will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Intraoperative remifentayl consumption (microgram) | peroperatively
  Total amount of remifentanyl during the Intraoperative period
Postoperative visual analog scale(1-10) | at the postoperative 1. hour
  the investigators aimed to compare postoperative visual analog scale of two groups.The visual pain scale is measured with a ruler from 0 to 10 cm. 0 indicates no pain 10 indicates severe pain
Rate of heart beat (beat/min) | During the anesthesia, It will be evaluated at 1 hour intervals.
  the investigators aimed to compare intraoperative pulse rate of two groups
Value of systolic blood pressure (mmHg) | During the anesthesia, It will be evaluated at 1 hour intervals.
  the investigators aimed to compare intraoperative systolic blood pressure of two groups
Rate of systemic inflammation index: SII (Systemic immune inflammatory index) is the formulation of the values of platelets, neutrophils and lymphocytes in peripheral blood as P X N / L = SII. | At the preoperative and postoperative time points
  the investigators aimed to compare postoperative systemic inflammation index of two groups.

SECONDARY OUTCOMES:
Amount of postoperative creatinine (mg/dl) | At the postoperative 24.hour
  the investigators aimed to compare postoperative creatine of two groups
Amount of postoperative urea (mg/L) | at the postoperative 24.hour
  It will be aimed to compare postoperative urea of two groups
incidence of death (percentage of ) | at postoperative 1.year
  the investigators aimed to compare postoperative mortality of two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)

REFERENCES:
- [Background] Walter CM, Lee CS, Moore DL, Abbasian N, Clay SJ, Mecoli MD, Olbrecht VA, Batra M, Ding L, Yang F, Nair M, Huq A, Simpson BE, Brown RL, Garcia VF, Chidambaran V. Retrospective study comparing outcomes of multimodal epidural and erector spinae catheter pain protocols after pectus surgery. J Pediatr Surg. 2023 Mar;58(3):397-404. doi: 10.1016/j.jpedsurg.2022.06.017. Epub 2022 Jul 6. PMID 35907711
- [Background] Putowski Z, Majewska K, Gruca K, Zimnoch A, Szczepanska A, Krzych LJ, Jablonska B, Mrowiec S. Intraoperative Hypotension and Its Association with Postoperative Acute Kidney Injury in Patients Undergoing Pancreaticoduodenectomy: A 5-Year, Single-Center, Retrospective Cohort Study. Med Sci Monit. 2023 Apr 11;29:e938945. doi: 10.12659/MSM.938945. PMID 37038338
- [Background] Viderman D, Tapinova K, Nabidollayeva F, Tankacheev R, Abdildin YG. Intravenous versus Epidural Routes of Patient-Controlled Analgesia in Abdominal Surgery: Systematic Review with Meta-Analysis. J Clin Med. 2022 May 5;11(9):2579. doi: 10.3390/jcm11092579. PMID 35566705
- [Background] Jipa M, Isac S, Klimko A, Simion-Cotorogea M, Martac C, Cobilinschi C, Droc G. Opioid-Sparing Analgesia Impacts the Perioperative Anesthetic Management in Major Abdominal Surgery. Medicina (Kaunas). 2022 Mar 28;58(4):487. doi: 10.3390/medicina58040487. PMID 35454326
- [Background] Nair A, Saxena P, Borkar N, Rangaiah M, Arora N, Mohanty PK. Erector spinae plane block for postoperative analgesia in cardiac surgeries- A systematic review and meta-analysis. Ann Card Anaesth. 2023 Jul-Sep;26(3):247-259. doi: 10.4103/aca.aca_148_22. PMID 37470522
- [Background] Zhang Y, Chong JH, Harky A. Enhanced recovery after cardiac surgery and its impact on outcomes: A systematic review. Perfusion. 2022 Mar;37(2):162-174. doi: 10.1177/0267659121988957. Epub 2021 Jan 19. PMID 33468017
- [Background] Chen Q, Ren S, Cui S, Huang J, Wang D, Li B, He Q, Lang R. Prognostic and recurrent significance of SII in patients with pancreatic head cancer undergoing pancreaticoduodenectomy. Front Oncol. 2023 May 22;13:1122811. doi: 10.3389/fonc.2023.1122811. eCollection 2023. PMID 37284203
- [Background] Canikli Adiguzel S, Akyurt D, Bahadir Altun H, Tulgar S, Ultan Ozgen G. Can Neutrophil-Lymphocyte Ratio, Platelet-Lymphocyte Ratio, or Systemic Immune Inflammation Index Be an Indicator of Postoperative Pain in Patients Undergoing Laparoscopic Cholecystectomy? Cureus. 2023 Jan 19;15(1):e33955. doi: 10.7759/cureus.33955. eCollection 2023 Jan. PMID 36820108